CLINICAL TRIAL: NCT07227714
Title: A Cluster-Randomized Trial Evaluating the Effect of Vision Centers on Access to Eye Care and Eye Health Outcomes in South Asia
Brief Title: Effect of Vision Centers on Access to Eye Care and Eye Health Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Seva Foundation (Other); Proctor Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 25-45086
Record Dates: First submitted 2025-11-10; First posted 2025-11-13 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Cataract Surgery; Eye Care; Glasses; Primary Eye Care; Vision Center; Eyecare Visits
Keywords: vision center; primary eye care; cataract surgery; glasses; glassess ownership; spectacle ownership; cluster-randomized trial; eyecare visits

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Survey data collectors and data analysts conducting the primary analyses will be masked. This will be achieved by not informing survey data collectors of arm assignment and by having an unmasked team member conceal arm assignment before primary analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate establishment of a vision center (Experimental): The intervention arm will include the establishment of a fixed vision center equipped with trained vision technicians to provide basic eye care services and referrals to higher care.
  Interventions: Other: Establishment of a vision center
- Delayed establishment of a vision center (No Intervention): The control arm will receive no intervention during the study period. The establishment of a vision center will occur after endline data collection, if hospital interest and resources remain adequate.

INTERVENTIONS:
Other: Establishment of a vision center — The establishment of a vision center includes building a fixed center, and equipping it with a trained vision technician to provide basic eye care services such as refractive error correction, spectacle dispensing, basic diagnosis for common conditions, as well as referrals for advanced care at base hospitals. The establishment of VCs will be actively publicized in the neighboring communities through promotion by local stakeholders, teachers, community workers, village leaders, health workers, and radio announcements prior to establishment. Additional outreach activities include posters and loudspeaker announcements in the communities the day before operations begin.
  Arms: Immediate establishment of a vision center

SUMMARY:
The goal of this clinical trial is to evaluate the effect of vision centers on access to eye care and eye health outcomes in South Asia. The main questions it aims to answer are:

1. Do vision centers increase visits to eyecare centers?
2. Do vision centers increase spectacle ownership and wearing?
3. Do vision centers improve visual acuity of the population?

Researchers will compare outcomes in communities randomized to have a vision center is established with communities randomized to delay establishment of a vision center. Outcomes will be assessed through population-based surveys at baseline and after two years as well as through hospital records collected throughout the study period.

DETAILED DESCRIPTION:
The vast majority of visual impairment and blindness is preventable or treatable with existing interventions. Nearly all of this burden is faced by those living in low- and middle-income countries. Access to eye care is a key challenge in these settings, particularly in rural and remote areas.

Vision centers (VCs) have been developed to increase access to primary eye care in such underserved settings. VCs typically involve establishment of a fixed center staffed by a mid-level ophthalmic technician who offers refraction, spectacles, diagnosis and treatment of basic eye conditions, and referrals for more complex care. VCs have become a common approach to increase access to care in many low- and middle-income country settings, yet little rigorous evidence exists on their impact on eye health in the communities they serve. A recent literature review was unable to identify randomized controlled trials on the impact of vision centers on eye health outcomes in real world settings. While the observational research that exists suggests VCs improve eye health in the communities they serve, the existing evidence is prone to bias.

The investigators propose a cluster-randomized trial to evaluate the effect of VCs on access to eye care and eye health outcomes in South Asia. The trial will leverage VCs planned by the Seva Foundation and partners Bangladesh, India, and Nepal and will monitor outcomes via population-based surveys and hospital network records over 2 years. The investigators expect to provide rigorous evidence on VC impact in real-world settings that can be used to influence programmatic decision making and policy.

ELIGIBILITY:
Inclusion Criteria:

* The catchment area of the proposed VC site is predominantly rural.
* The proposed VC site is located within 20-100 km of the base hospital.
* There are no major primary eye care services within 10 km of the proposed site.
* Care at sites randomized to establish VCs immediately is accessible to anyone.

Exclusion Criteria:

* Sites located in non-rural or urban catchment areas.
* Sites outside the 20-100 km distance range from the base hospital.
* Sites with existing major primary eye care services within a 10 km radius.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of eyecare visits | 1 year
  The primary outcome is the prevalence of eyecare visits completed in the past one year, defined for each cluster as the number of individuals having completed at least one visit in the past year divided by the total number of individuals surveyed.

SECONDARY OUTCOMES:
Total number of visits to any eyecare provider | 1 year
  Total number of visits to any eyecare provider within the past 12 months as reported during the survey (overall and among those with visual impairment).
Prevalence of current spectacle ownership | 2 years.
  Prevalence of current spectacle ownership assessed during the population-based survey among all age groups.
Effective refractive error coverage | 2 years
  Defined as the proportion of survey participants with met need for refractive error correction with good quality vision of 6/12 or better in the better seeing eye divided by the total number of people in need (met need + undermet need + unmet need).
Prevalence of spectacle wearing | 2 years
  Prevalence of spectacle wearing as assessed during the survey among all age groups.
Mean presenting and pinhole visual acuity | 2 years
  Mean presenting and pinhole visual acuity (logMAR) as assessed during the survey among adults 50 years and older, among children younger than 18 years, and among all ages.
Prevalence of visual impairment | 2 years
  Visual impairment is defined as presenting visual acuity worse than logMAR 0.54 in the better-seeing eye as assessed during the population-based survey, for adults aged 50 years and older, children younger than 18 years, and all ages.
Prevalence of blindness | 2 years
  Blindness is defined as presenting visual acuity worse than logMAR 1.30 in the better-seeing eye as assessed during the population-based survey, for adults aged 50 years and older, children younger than 18 years, and all ages.
Number of eye surgeries | 2 years
  Number of eye surgeries as reported by participants during the survey among adults 50 years and older.
Prevalence of other ocular diagnoses and treatment/procedures | 2 years
  Prevalence of other ocular diagnoses and treatment/procedures assessed during the population-based survey among all age groups.
Prevalence of employment | 2 years
  Prevalence of employment as assessed during the population-based survey among adults 18 years and older.
Mean annual household income | 2 years
  Mean annual household income as assessed during the population-based survey, converted to a common currency (USD) and adjusted for purchasing power parity (international dollars).
Prevalence of individuals with caregiving responsibilities for visually impaired household members | 2 years
  Prevalence of individuals with caregiving responsibilities for visually impaired household members assessed during the population-based survey.
Total number of network visits | 2 years
  Captured from passive surveillance
Cause-specific number of network visits | 2 years
  Number of network visits for specific causes including cataract, refractive error, diabetic retinopathy, glaucoma, and age-related macular degeneration, captured by passive surveillance of hospital data.
Number of cataract surgeries performed | 2 years
  Captured from passive surveillance
Cost of vision center implementation | 2 years
  Program costs of vision center implementation will be measured, with cost categories including personnel, equipment, supplies, training, transportation, and infrastructure.
Cost effectiveness of vision center | 2 years
  The cost effectiveness will be calculated as the incremental cost per additional cataract surgery performed in the intervention arm. Incremental cost-effectiveness ratios (ICERs) will be calculated using program costs and cataract surgeries enumerated from the hospitals during the study time period.

CONTACTS AND LOCATIONS:
Overall Officials: Kieran O'Brien, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified cluster-level data will be shared publicly via osf.io
Supporting Information: Study Protocol
Time Frame: Within 6 months after the study ends.
Access Criteria: General public
URL: https://osf.io/

REFERENCES:
- [Background] Khanna RC, Sabherwal S, Sil A, Gowth M, Dole K, Kuyyadiyil S, Chase H. Primary eye care in India - The vision center model. Indian J Ophthalmol. 2020 Feb;68(2):333-339. doi: 10.4103/ijo.IJO_118_19. PMID 31957722
- [Background] Rao GN, Khanna RC, Athota SM, Rajshekar V, Rani PK. Integrated model of primary and secondary eye care for underserved rural areas: the L V Prasad Eye Institute experience. Indian J Ophthalmol. 2012 Sep-Oct;60(5):396-400. doi: 10.4103/0301-4738.100533. PMID 22944748
- [Background] Misra V, Vashist P, Malhotra S, Gupta SK. Models for primary eye care services in India. Indian J Community Med. 2015 Apr-Jun;40(2):79-84. doi: 10.4103/0970-0218.153868. PMID 25861167
- [Background] Vision Loss Expert Group of the Global Burden of Disease Study; GBD 2019 Blindness and Vision Impairment Collaborators. Global estimates on the number of people blind or visually impaired by cataract: a meta-analysis from 2000 to 2020. Eye (Lond). 2024 Aug;38(11):2156-2172. doi: 10.1038/s41433-024-02961-1. PMID 38461217
- [Background] Vision Loss Expert Group of the Global Burden of Disease Study; GBD 2019 Blindness and Vision Impairment Collaborators. Global estimates on the number of people blind or visually impaired by Uncorrected Refractive Error: a meta-analysis from 2000 to 2020. Eye (Lond). 2024 Aug;38(11):2083-2101. doi: 10.1038/s41433-024-03106-0. Epub 2024 Jul 4. PMID 38965322
- [Background] GBD 2019 Blindness and Vision Impairment Collaborators; Vision Loss Expert Group of the Global Burden of Disease Study. Trends in prevalence of blindness and distance and near vision impairment over 30 years: an analysis for the Global Burden of Disease Study. Lancet Glob Health. 2021 Feb;9(2):e130-e143. doi: 10.1016/S2214-109X(20)30425-3. Epub 2020 Dec 1. PMID 33275950
- [Background] GBD 2019 Blindness and Vision Impairment Collaborators; Vision Loss Expert Group of the Global Burden of Disease Study. Causes of blindness and vision impairment in 2020 and trends over 30 years, and prevalence of avoidable blindness in relation to VISION 2020: the Right to Sight: an analysis for the Global Burden of Disease Study. Lancet Glob Health. 2021 Feb;9(2):e144-e160. doi: 10.1016/S2214-109X(20)30489-7. Epub 2020 Dec 1. PMID 33275949
- [Background] Burton MJ, Ramke J, Marques AP, Bourne RRA, Congdon N, Jones I, Ah Tong BAM, Arunga S, Bachani D, Bascaran C, Bastawrous A, Blanchet K, Braithwaite T, Buchan JC, Cairns J, Cama A, Chagunda M, Chuluunkhuu C, Cooper A, Crofts-Lawrence J, Dean WH, Denniston AK, Ehrlich JR, Emerson PM, Evans JR, Frick KD, Friedman DS, Furtado JM, Gichangi MM, Gichuhi S, Gilbert SS, Gurung R, Habtamu E, Holland P, Jonas JB, Keane PA, Keay L, Khanna RC, Khaw PT, Kuper H, Kyari F, Lansingh VC, Mactaggart I, Mafwiri MM, Mathenge W, McCormick I, Morjaria P, Mowatt L, Muirhead D, Murthy GVS, Mwangi N, Patel DB, Peto T, Qureshi BM, Salomao SR, Sarah V, Shilio BR, Solomon AW, Swenor BK, Taylor HR, Wang N, Webson A, West SK, Wong TY, Wormald R, Yasmin S, Yusufu M, Silva JC, Resnikoff S, Ravilla T, Gilbert CE, Foster A, Faal HB. The Lancet Global Health Commission on Global Eye Health: vision beyond 2020. Lancet Glob Health. 2021 Apr;9(4):e489-e551. doi: 10.1016/S2214-109X(20)30488-5. Epub 2021 Feb 16. No abstract available. PMID 33607016